CLINICAL TRIAL: NCT01506882
Title: An Open-label, Randomized, Multicenter Study to Evaluate the Efficacy and Safety of Levetiracetam Used as Monotherapy in Newly or Recently Diagnosed Epilepsy Patients Aged Older Than or Equal to 16 Years With Partial Seizures
Brief Title: An Open Label Study of Levetiracetam Monotherapy in Patients With Newly Diagnosed Focal Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N01375; 2014-004377-16 (EudraCT Number)
Record Dates: First submitted 2012-01-05; First posted 2012-01-10 (Estimated); Results first posted 2014-10-13 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-11

CONDITIONS: Epilepsy; Partial Onset Seizures
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam 1000 mg/day to 2000 mg/day group (Experimental): Subjects in the LEV 1000 mg/day to 2000 mg/day group receive the initial dose of LEV 1000 mg/day for the 1- week Stabilization Period and enter the Evaluation Period. Unless a seizure occurs during the Evaluation Period, the subjects will continue LEV 1000 mg/day for 26 weeks. If a seizure occurs during the Evaluation Period, the dose will be increased to 2000 mg/day and a restart of stabilization on LEV 2000 mg/day for 1 week is required prior to restarting the 26-weeks Evaluation Period on LEV 2000 mg/day.
  The LEV dose could be decreased as a fallback option at the investigator's discretion, if the subject did not tolerate the LEV dosage, as evidenced by the development of an AE. The fallback option was permitted to be performed once for subjects on LEV 2000 mg/day at any time during the restarted Stabilization Period (SP), restarted Evaluation Period (EP), or Maintenance Period (MP), as well as for subjects on LEV 3000 mg/day at any time during the SP, EP, or MP.
  Interventions: Drug: Levetiracetam (LEV)
- Levetiracetam 3000 mg/day group (Experimental): Unless a seizure occurs, the subjects in this arm will continue LEV 3000 mg/day for 26 weeks. Subjects in the LEV 3000 mg/day group undergo a 4-week Up-Titration Period prior to the 1-week Stabilization Period.
  They receive 1000 mg/day for 2 weeks and 2000 mg/day for 2 weeks during the Up-Titration Period and LEV 3000 mg/day for 1 week during the Stabilization Period.
  The LEV dose could be decreased as a fallback option at the investigator's discretion, if the subject did not tolerate the LEV dosage, as evidenced by the development of an AE. The fallback option was permitted to be performed once for subjects on LEV 2000 mg/day at any time during the restarted Stabilization Period (SP), restarted Evaluation Period (EP), or Maintenance Period (MP), as well as for subjects on LEV 3000 mg/day at any time during the SP, EP, or MP.
  Interventions: Drug: Levetiracetam (LEV)

INTERVENTIONS:
Drug: Levetiracetam (LEV) — * Active Substance: Levetiracetam
  * Pharmaceutical Form: Film-coated tablet
  * Concentration: LEV 250 mg, LEV 500 mg
  * Frequency: Twice daily
  * Route of Administration: Oral use
  Other Names: Keppra; E Keppra

SUMMARY:
The purpose of this study is to evaluate the efficacy of Levetiracetam (LEV) used as monotherapy, with efficacy measured as 6-month seizure freedom at the last evaluated dose in the LEV 1000 mg/day to 2000 mg/day group, in newly or recently diagnosed epilepsy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and aged ≥ 16 years at Visit 1
* Subjects with newly or recently diagnosed Epilepsy having experienced unprovoked Partial Seizures (IA, IB, IC), that are classifiable according to the International League Against Epilepsy (ILAE) classification of Epileptic Seizures
* Subjects with at least 2 unprovoked seizures separated by a minimum of 48 hours in the year prior to Visit 1, of which, at least 1 unprovoked seizure occurred in the 3 months prior to Visit 1
* Minimum body weight of 40 kg at Visit 1

Exclusion Criteria:

* Subject has a history or presence of seizure types other than partial (IA, IB, IC)
* Subject has an experience of any type of brain surgery in the consecutive 2 years prior to Visit 1
* Subject has a history or presence of known Pseudo-Seizures
* Subject has been treated for Epilepsy with any Antiepileptic Drug (AED) within the 6 months prior to Visit 1. However, acute and sub-acute seizure treatments are accepted for a maximum use of 2 weeks, if the treatments are stopped for the week prior to Visit 1
* Subject has a known clinically significant acute or chronic illness, such as but not restricted to: cardiac, renal, hepatic dysfunction, endocrinological, or psychiatric illness, and that may impair reliable participation in the study or necessitate the use of medication not allowed by the protocol

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-12; Primary Completion 2013-10 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (27):
- Japan (27):
  - 19, Aomori
  - 33, Asaka
  - 21, Daitō
  - 12, Fujisawa
  - 14, Hamamatsu
  - 11, Himeji
  - 30, Hirosaki
  - 8, Kagoshima
  - 20, Kamakura
  - 17, Kawasaki
  - 3, Kitakyushu
  - 26, Kodaira
  - 9, Kokubunji
  - 32, Kyoto
  - 25, Miyakonojō
  - 5, Nagoya Aichi
  - 4, Nara
  - 22, Okayama
  - 15, Osaka
  - 27, Osaka
  - 13, Saitama
  - 1, Sakai
  - 29, Sapporo
  - 24, Sayama
  - 2, Toyonaka
  - 7, Ube
  - 18, Yamagata

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study started to enroll subjects in December 2011 in order to end up with 27 centers with enrolled subjects in Japan.
Pre-assignment Details: Participant Flow refers to the Randomized Set (RS). RS consists of all subjects who were randomized to the study groups.
Groups:
- Levetiracetam 1000 mg/Day to 2000 mg/Day Group: * Formulation: Tablet
  * Strength: LEV 250 mg, LEV 500 mg
  * Dosage: First study dose is 1000 mg/day and if a seizure occurs, the dose will be increased to 2000 mg/day. Max dose in the Follow Up Period is 3000 mg/day.
  * Frequency: Twice daily
- Levetiracetam 3000 mg/Day Group: * Formulation: Tablet
  * Strength: LEV 250 mg, LEV 500 mg
  * Dosage: 1000 mg/day for first two weeks, then 2000 mg/day for two weeks then 3000 mg/day by the end of the trial.
  * Frequency: Twice daily
Period: Overall Study
Arm/Group | Levetiracetam 1000 mg/Day to 2000 mg/Day Group | Levetiracetam 3000 mg/Day Group
Started | 61 | 10
Completed | 39 | 3
Not Completed | 22 | 7
Not completed — Lack of Efficacy | 4 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 9 | 3
Not completed — SAE, non-fatal | 2 | 0
Not completed — AE, non-serious non-fatal | 3 | 1
Not completed — SAE,non-fatal+AE,non-serious non-fatal | 1 | 0
Not completed — Other Reason | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set (SS). SS consists of all subjects in the Enrolled Set, who received at least 1 dose of the Investigational Medicinal Product (IMP).
Arm/Group | Levetiracetam 1000 mg/Day to 2000 mg/Day Group | Levetiracetam 3000 mg/Day Group | Total Title
Number analyzed (Participants) | 61 | 10 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 1 | 11
  Between 18 and 65 years | 45 | 8 | 53
  >=65 years | 6 | 1 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (18.0) | 37.0 (18.6) | 36.5 (17.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 4 | 38
  Male | 27 | 6 | 33
Region of Enrollment [Number; unit: participants]
  Japan | 61 | 10 | 71
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 58.98 (12.30) | 62.58 (15.11) | 59.48 (12.67)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 161.96 (8.77) | 166.07 (10.21) | 162.54 (9.02)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects in the Levetiracetam (LEV) 1000 mg/Day to 2000 mg/Day Group Who Are Seizure Free for 26 Consecutive Weeks of Treatment During the Evaluation Period
Description: A subject was considered seizure free, if no seizure occurred during the 6 consecutive months (26 weeks) in the Evaluation Period. If one of the following occurred, the subject was not considered seizure free:
  * A documented seizure during 6 consecutive months of the Evaluation Analysis Period
  * Subject discontinued the study prematurely during the Evaluation Analysis Period
  * Missing Seizure Count Case Report Forms (CRFs) prior to completing the Evaluation Analysis Period.
Time Frame: From the end of the 1-week Stabilization Period over the 26-weeks Evaluation Period
Population: Data for the primary outcome measure refer to the Full Analysis Set (FAS). FAS includes all subjects in the Safety Set who had at least 1 treatment day in the Evaluation Period. This means that subjects in LEV 1000 to 2000 mg/day group had to have at least 1 treatment day in the Evaluation Period on their final evaluated dose.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Levetiracetam 1000 mg/Day to 2000 mg/Day Group
Number analyzed (Participants) | 61
percentage of participants | 73.8 [60.9 to 84.2]
Statistical Analysis 1: Comparison: Levetiracetam 1000 mg/Day to 2000 mg/Day Group; The primary efficacy variable was to be calculated as the proportion p=n/N of subjects (n) staying seizure free for 6 months out of the total number of subjects (N). For this proportion p, an exact 2-sided 95% confidence interval (CI) was computed based on the F distribution. The hypothesis H0: p=0.4 was to be formally rejected in favor of H1: p>0.4, if the lower confidence limit for p was greater than 0.4; Test type: Superiority or Other; Percent = 73.8, 95% CI 2-sided [60.9 to 84.2]

2. Secondary Outcome: Percentage of Subjects in the Levetiracetam (LEV) 1000 mg/Day to 2000 mg/Day Group Who Are Seizure Free for 52 Consecutive Weeks of Treatment During the Evaluation Period and the Maintenance Period
Description: Subjects who complete the 26-weeks Evaluation Period without having a seizure will continue receiving the same dose of LEV as in the Evaluation Period during the 26-weeks Maintenance Period unless a seizure occurs.
Time Frame: From entry in the 26-weeks Evaluation Period to the end of the 26-weeks Maintenance Period
Population: Data for this secondary outcome measure refer to the Full Analysis Set (FAS). FAS includes all subjects in the Safety Set who had at least 1 treatment day in the Evaluation Period. This means that subjects in LEV 1000 to 2000 mg/day group had to have at least 1 treatment day in the Evaluation Period on their final evaluated dose.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Full Analysis Set (LEV 1000 mg/Day to 2000 mg/Day Group): FAS includes all subjects in the Safety Set who had at least 1 treatment day in the Evaluation Period. This means that subjects in LEV 1000 to 2000 mg/day group had to have at least 1 treatment day in the Evaluation Period on their final evaluated dose.
  * Formulation: Tablet
  * Strength: LEV 250 mg, LEV 500 mg
  * Dosage: First study dose is 1000 mg/day and if a seizure occurs, the dose will be increased to 2000 mg/day. Max dose in the Follow Up Period is 3000 mg/day.
  * Frequency: Twice daily
Arm/Group | Full Analysis Set (LEV 1000 mg/Day to 2000 mg/Day Group)
Number analyzed (Participants) | 61
percentage of participants | 59.0 [45.7 to 71.4]

3. Secondary Outcome: Percentage of Subjects in the Levetiracetam (LEV) 3000 mg/Day Group Who Are Seizure Free for 26 Consecutive Weeks of Treatment During the Evaluation Period
Description: as for outcome 1
Time Frame: From the end of the 1-week Stabilization Period over the 26-weeks Evaluation Period
Population: Data for this secondary outcome measure refer to the Full Analysis Set (FAS). FAS includes all subjects in the Safety Set who had at least 1 treatment day in the Evaluation Period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Levetiracetam 3000 mg/Day Group
Number analyzed (Participants) | 9
percentage of participants | 22.2 [2.8 to 60.0]

4. Secondary Outcome: Percentage of Subjects in the Levetiracetam (LEV) 3000 mg/Day Group Who Are Seizure Free for 52 Consecutive Weeks of Treatment During the Evaluation Period and the Maintenance Period
Description: Subjects who complete the 26-weeks Evaluation Period without having a seizure will continue receiving LEV 3000 mg/day during the 26-weeks Maintenance Period unless a seizure occurs.
Time Frame: From entry in the 26-weeks Evaluation Period to the end of the 26-weeks Maintenance Period
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Full Analysis Set (LEV 3000 mg/Day Group): FAS includes all subjects in the Safety Set who had at least 1 treatment day in the Evaluation Period. This means that subjects in LEV 1000 to 2000 mg/day group had to have at least 1 treatment day in the Evaluation Period on their final evaluated dose.
  * Formulation: Tablet
  * Strength: LEV 250 mg, LEV 500 mg
  * Dosage: 1000 mg/day for first two weeks, then 2000 mg/day for two weeks then 3000 mg/day by the end of the trial.
  * Frequency: Twice daily
Arm/Group | Full Analysis Set (LEV 3000 mg/Day Group)
Number analyzed (Participants) | 9
percentage of participants | 11.1 [0.3 to 48.2]

5. Secondary Outcome: Time to First Seizure at the Last Evaluated Dose in Subjects in the Levetiracetam (LEV) 1000 mg/Day to 2000 mg/Day Group
Description: Time was measured from first day of last evaluated dose. Seizures during Stabilization were not considered.
  The Median time to first seizure will be estimated from the Kaplan-Meier curve.
Time Frame: During Evaluation, Maintenance and Safety Follow Up Period after 1-week Stabilization Period, assessed up to 1 year
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Full Analysis Set (LEV 1000 mg/Day to 2000 mg/Day Group)
Number analyzed (Participants) | 61
days | NA [359 to NA] — values not estimable due to small number of events

6. Secondary Outcome: Time to Withdrawal at the Last Evaluated Dose in Subjects in the Levetiracetam (LEV) 1000 mg/Day to 2000 mg/Day Group
Description: Median time to withdrawal will be estimated from the Kaplan-Meier curve.
Time Frame: During 1-week Stabilization Period, Evaluation, Maintenance and Safety Follow Up Period, assessed up to 1 year
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Full Analysis Set (LEV 1000 mg/Day to 2000 mg/Day Group)
Number analyzed (Participants) | 61
days | NA [NA to NA] — values not estimable due to small number of events

7. Secondary Outcome: Time to First Seizure in Subjects in the Levetiracetam (LEV) 3000 mg/Day Group
Description: as for outcome 5
Time Frame: During Evaluation, Maintenance and Safety Follow Up Period after 1-week Stabilization Period, assessed up to 1 year
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Full Analysis Set (LEV 3000 mg/Day Group)
Number analyzed (Participants) | 9
days | 106 [9 to NA] — value not estimable due to small number of events

8. Secondary Outcome: Time to Withdrawal in Subjects in the Levetiracetam (LEV) 3000 mg/Day Group
Description: Median time to withdrawal will be estimated from the Kaplan-Meier curve.
Time Frame: During 1-week Stabilization Period, Evaluation, Maintenance and Safety Follow Up Period, assessed up to 1 year
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Levetiracetam 3000 mg/Day Group
Number analyzed (Participants) | 9
days | 91 [21 to 197]

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events were collected from Screening (Week 0) over the Evaluation and Maintenance Period (Week 4 to Week 53) until the last Follow-up Visit or Withdrawal Visit.
Description: Adverse Events refer to the Safety Set, which includes all subjects in the Enrolled Set who received at least 1 dose of the Investigational Medicinal Product.
Arm/Group | Levetiracetam 1000 mg/Day to 2000 mg/Day Group | Levetiracetam 3000 mg/Day Group
Serious Adverse Events (participants affected / at risk) | 8/61 | 2/10
Other Adverse Events (participants affected / at risk) | 58/61 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam 1000 mg/Day to 2000 mg/Day Group (N=61) | Levetiracetam 3000 mg/Day Group (N=10)
Irritability (General disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Kaposi's varicelliform eruption (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 3 (3) | 0 (0)
Postictal state (Nervous system disorders) | 2 (2) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Postictal psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (2) | 0 (0)
Meniscus removal (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam 1000 mg/Day to 2000 mg/Day Group (N=61) | Levetiracetam 3000 mg/Day Group (N=10)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 8 (18) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (14) | 1 (1)
Dental caries (Gastrointestinal disorders) | 6 (7) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 4 (17) | 0 (0)
Gastritis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (5) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 12 (13) | 0 (0)
Pyrexia (General disorders) | 5 (6) | 1 (2)
Nasopharyngitis (Infections and infestations) | 47 (155) | 4 (7)
Influenza (Infections and infestations) | 7 (8) | 0 (0)
Cystitis (Infections and infestations) | 4 (5) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 5 (6) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Weight increased (Investigations) | 2 (2) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 1 (1)
Urine ketone body present (Investigations) | 2 (2) | 1 (1)
Blood urine present (Investigations) | 1 (1) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 25 (32) | 2 (2)
Headache (Nervous system disorders) | 10 (14) | 1 (1)
Dizziness (Nervous system disorders) | 8 (9) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 1 (1)
Amnestic disorder (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Ketonuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 5 (8) | 0 (0)
Acquired phimosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days